CLINICAL TRIAL: NCT05299931
Title: An Open-Label Extension and Long-term Efficacy and Safety Monitoring Study of Patients with Crohn's Disease Previously Included in the Loss of RESponse to Ustekinumab Treated by Dose Escalation Study (REScUE-OLE)
Brief Title: An Open-Label Extension and Long-term Efficacy and Safety Monitoring Study of Patients with Crohn's Disease Previously Included in the Loss of RESponse to Ustekinumab Treated by Dose Escalation Study
Acronym: REScUE-OLE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Belgian Inflammatory Bowel Disease Research and Development (BIRD) VZW (Other)
Collaborators: Janssen Cilag N.V./S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIRD2020001
Record Dates: First submitted 2022-02-09; First posted 2022-03-29 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease
Keywords: ustekinumab
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subcutaneous (SC) ustekinumab every 8 weeks (Q8w) (Other): Patients previously enrolled to the ustekinumab 90 mg SC Q8w-arm will continue ustekinumab 90 mg SC Q8w if they are "Q8w responders" at the end of REScUE
  Patients treated with a OLE treatment regimen of ustekinumab 90 mg SC Q8w will be able to cross-over to a OLE treatment regimen of ustekinumab 90 mg SC Q4w if they meet the criteria of CD worsening at week 12 or at any timepoint beyond week 12 after entering REScUE-OLE
  Interventions: Drug: Ustekinumab
- Subcutaneous (SC) ustekinumab every 4 weeks (Q4w) (Other): Patients previously enrolled to the ustekinumab 90 mg SC Q8w-arm will switch to ustekinumab 90 mg SC Q4w ("Cross-over") if they are "Q8w non-responders" at the end of REScUE OR Patients previously enrolled to the ustekinumab 90 mg SC Q4w-arm will continue ustekinumab 90 mg SC Q4w if they are "Q4w responders" at the end of REScUE
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — dose escalation from every 8 weeks to every 4 weeks only in arm 2
  Other Names: dose escalation only in arm 2

SUMMARY:
The aim of the study is to assess the long-term efficacy and safety of a ustekinumab 90mg subcutaneous (SC) every 4 weeks (Q4w) regimen in patients with Crohn's disease previously enrolled in the REScUE study (NCT04245215) because of secondary loss of response to a ustekinumab 90mg SC every 8 weeks (Q8w) regimen.

DETAILED DESCRIPTION:
The study is a prospective, open-label study only enrolling patients that were previously included in the REScUE study (n=max. 108; NCT04245215) and that terminated that study at week 48. Patients will undergo most necessary examinations, including endoscopy, as part of the Week 48 visit of the REScUE study and those should therefore not be repeated as part of Week 0 visit of the REScUE-OLE study (W0 REScUE-OLE = W48 REScUE). The FACIT-Fatigue scale and the additional laboratory evaluations (serum creatinine, ALT, AST and conjugated bilirubin) are the only examinations that are not foreseen at the end of the REScUE study at week 48. During the 4-week period following the start of REScUE-OLE (= end of REScuE at Week 48), collection and monitoring of the patient's data within the REScUE study will first be finalized, after which unblinding takes place. Depending on the final outcome and treatment of the patient in REScUE ("Q8w responders", "Q8w non-responders", "Q4w responders"), the OLE treatment regimen will be decided as follows:

1. Patients previously enrolled to the ustekinumab 90 mg SC Q8w-arm will continue ustekinumab 90 mg SC Q8w if they are "Q8w responders" at the end of REScUE, defined by the following criteria:

   * Concomitant steroid use <= 20 mg prednisone equivalents (budesonide <=6 mg; beclomethasone dipropionaat <= 5 mg) for at least 28 days before the end of REScUE at week 48 AND
   * Clinical remission (defined as average AP <=1 and average SF <=3) OR clinical response (defined as a drop of at least 50% in average AP and/or a drop of at least 50% in average SF as compared to REScUE baseline, and both average AP and SF no worse than REScUE baseline) AND
   * Endoscopic remission (defined as a total SES-CD <5) OR endoscopic response (defined as a drop of at least 50% in total SES-CD score as compared to REScUE baseline)
2. Patients previously enrolled to the ustekinumab 90 mg SC Q8w-arm will switch to ustekinumab 90 mg SC Q4w ("Cross-over") if they are "Q8w non-responders" at the end of REScUE, defined as failing to meet the criteria for continuation of ustekinumab 90 mg SC Q8w as described above (in 1).
3. Patients previously enrolled to the ustekinumab 90 mg SC Q4w-arm will continue ustekinumab 90 mg SC Q4w if they are "Q4w responders" at the end of REScUE, defined by the following criteria:

   * Concomitant steroid use <=20 mg prednisone equivalents (budesonide <=6 mg; beclomethasone dipropionaat <=5 mg) for at least 28 days before the end of REScUE at week 48 AND
   * Clinical remission (defined as average AP <=1 and average SF <=3) OR clinical response (defined as a drop of at least 50% in average AP and/or a drop of at least 50% in average SF as compared to REScUE baseline, and both average AP and SF no worse than REScUE baseline) AND
   * Endoscopic remission (defined as a total SES-CD <5) OR endoscopic response (defined as a drop of at least 50% in total SES-CD score as compared to REScUE baseline)
4. Patients previously enrolled to the ustekinumab 90 mg SC Q4w-arm will be excluded from continuation of treatment within REScUE-OLE ("Screen failure") if they are "Q4w non-responders" at the end of REScUE, defined as failing to meet the criteria for continuation of ustekinumab 90 mg SC Q4w as described above (in 3).

The consecutive CD treatment after REScUE-OLE cessation is at the discretion of the treating physician.

During the REScUE-OLE study, patients will have on-site, scheduled visits at 5 different timepoints. At each of these visits, the following study procedures will take place: registration of current (CD and non-CD) treatment, assessments of (serious) adverse events, disease activity assessment (PRO-2), physical examination, weight assessment, assessment of vital signs (blood pressure and pulse), laboratory evaluation (including CRP, haemoglobin, thrombocytes, serum albumin, serum creatinine, ALT, AST, conjugated bilirubin, and FC), patient diary review and instruction, and administration of commercially available ustekinumab 90 mg SC. At week 56 and at the end of the study at week 112, these study procedures will be complemented with pharmacokinetic sampling, an ileocolonoscopy and a monitoring of quality-of-life, work and productivity impairment and fatigue, using dedicated questionnaires. For all visits, a window of maximum 7 days is authorized. In between on-site visits, the administration of the medication is allowed off-site, following the schedule of the OLE treatment arm in which they are allocated. This can either be done by self-administration, for patients who have been trained to self-administer, or by a qualified medical professional.

Steroid use at the start and during the study is possible, but a strict tapering regimen is mandatory. Dose-escalation or (re-)initiation of steroids is allowed for a maximum of two times during the study period, with at least 6 months between the first and the second steroid dose-escalation/(re-)initiation. Patients treated with ustekinumab 90 mg SC Q8w will be able to cross-over to a ustekinumab 90 mg SC Q4w regimen if they meet the criteria of CD worsening at week 12 or at any timepoint beyond week 12 after entering REScUE-OLE. Patients treated with a OLE treatment regimen of ustekinumab 90 mg SC Q4w will stop the REScUE-OLE study and discontinue ustekinumab within the REScUE-OLE study, if they meet the criteria of CD worsening at two different timepoints (separated by at least 4 weeks) beyond week 12 after initiation of this OLE treatment regimen.

Primary endpoint of the REScUE-OLE study (sustained steroid-free clinical remission) will be assessed at week 112.

ELIGIBILITY:
Inclusion Criteria:

1. Previous inclusion in the REScUE study and having reached the end of this study at week 48.
2. Adequate contraception in females of reproductive age (oral, transdermal, injectable contraception, intra-uterine device, sterilisation or barrier method). Adequate contraception in males (sterilization or barrier method) if his female partner is of reproductive age.
3. Have the capacity to understand and sign an informed consent form.
4. Be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Patients previously enrolled to the ustekinumab 90 mg SC Q4w-arm during REScUE who were on concomitant steroid use >20 mg prednisone equivalents (budesonide >6 mg; beclomethasone dipropionaat >5 mg) at any time point in the last 28 days before the end of REScUE at week 48.
2. Patients previously enrolled to the ustekinumab 90 mg SC Q4w-arm during REScUE that did not reach the following criteria at the end of REScUE at week 48:

   * Clinical remission (defined as average AP<=1 and average SF<=3) OR clinical response (defined as a drop of at least 50% in average AP and/or a drop of at least 50% in average SF as compared to REScUE baseline, and both average AP and SF no worse than REScUE baseline) AND
   * Endoscopic remission (defined as a total SES-CD <5) OR endoscopic response (defined as a drop of at least 50% in total SES-CD score as compared to REScUE baseline)
3. Patients who developed an anaphylactic or severe allergic reaction to study medication during REScUE.
4. Patients with any of the following laboratory tests at W0 of the REScUE-OLE study :

   * Hemoglobin level <8.5 g/dL
   * Platelets level <100.000 /mm3
   * Serum creatinine level ≥1.7 mg/dL
   * AST and ALT level >3 times the upper limit of normal range
   * Direct (conjugated) bilirubin level ≥3.0 mg/dL
5. Patients with an ongoing treatment with another concomitant biological (vedolizumab, anti-TNF), a JAK-inhibitor or any investigational product for the treatment of Crohn's disease at the end of REScUE at week 48.
6. Patients who experience or have an ongoing infection event confirmed by positive stool or blood testing (including gastrointestinal pathogens, tuberculosis, HIV, hepatitis B, hepatitis C) should not initiate REScUE-OLE until (i) this event has completely resolved as shown by the termination of treatment with anti-infective medication, or (ii) this event is considered to be in stable remission under anti-infective medication in case of HIV, hepatitis B and hepatitis C.
7. Patients with an impassable stenosis even after attempt of endoscopic balloon dilatation.
8. Patients with an intra-abdominal abscess, or patients with an intra-anal abscess without adequate drainage by e.g. a seton placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in both treatment arms in steroid-free clinical remission | Week 56
  Proportion of patients in both treatment arms in steroid-free clinical remission (PRO-2 remission: average AP <=1 and average SF <=3 without any steroid use in the previous 28 days) at both week 56 and week 112 of the study (sustained steroid-free clinical remission).
Proportion of patients in both treatment arms in steroid-free clinical remission | Week 112
  Proportion of patients in both treatment arms in steroid-free clinical remission (PRO-2 remission: average AP <=1 and average SF <=3 without any steroid use in the previous 28 days) at both week 56 and week 112 of the study (sustained steroid-free clinical remission).

SECONDARY OUTCOMES:
Incidence and severity of adverse events in both treatment arms. | week 112
Time to CD worsening in both treatment arms | week 112
Proportion of patients in both treatment arms in steroid-free clinical remission (PRO-2 remission: average AP <=1 and average SF <=3 without any steroid use in the previous 28 days) at week 56 of the study. | Week 56
Proportion of patients in both treatment arms in steroid-free clinical remission (PRO-2 remission: average AP <=1 and average SF <=3 without any steroid use in the previous 28 days) at week 112 of the study. | Week 112
Proportion of patients previously enrolled to UST 90 mg SC Q8w-arm during REScUE who needed dose optimization to ustekinumab 90 mg SC Q4w at the start or during REScUE-OLE (<=week 100), and that reached steroid-free clinical remission at week 112. | Week 112
  Proportion of patients previously enrolled to the ustekinumab (UST) 90 mg SC Q8w-arm during REScUE who needed dose optimization to ustekinumab 90 mg SC Q4w at the start or during REScUE-OLE (<=week 100), and that reached steroid-free clinical remission (PRO-2 remission: average AP <=1 and average SF <=3 without any steroid use in the previous 28 days) at week 112.
Proportion of patients in both treatment arms in clinical remission (PRO-2 remission: average AP <=1 and average SF <=3) at week 56 of the study (sustained clinical remission). | Week 56
Proportion of patients in both treatment arms in clinical remission (PRO-2 remission: average AP <=1 and average SF <=3) at week 56 of the study. | Week 112
Proportion of patients previously enrolled to the ustekinumab 90 mg SC Q8w-arm during REScUE who needed dose optimization to ustekinumab 90 mg SC Q4w at the start or during REScUE-OLE (<=week 100), and that reached clinical remission at week 112. | Week 112
  Proportion of patients previously enrolled to the ustekinumab 90 mg SC Q8w-arm during REScUE who needed dose optimization to ustekinumab 90 mg SC Q4w at the start or during REScUE-OLE (<=week 100), and that reached clinical remission (PRO-2 remission: average AP <=1 and average SF <=3) at week 112.
Proportion of patients in both treatment arms with biomarker remission (CRP <5 mg/L and FC <=250 ug/g) at week 56 of the study. | Week 56
Proportion of patients in both treatment arms with biomarker remission (CRP <5 mg/L and FC <=250 ug/g) at week 112 of the study. | Week 112
Proportion of patients previously enrolled to the ustekinumab 90 mg SC Q8w-arm during REScUE who needed dose optimization to ustekinumab 90 mg SC Q4w at the start or during REScUE-OLE (<=week 100), and that reached biomarker remission at week 112. | Week 112
  Proportion of patients previously enrolled to the ustekinumab 90 mg SC Q8w-arm during REScUE who needed dose optimization to ustekinumab 90 mg SC Q4w at the start or during REScUE-OLE (<=week 100), and that reached biomarker remission (CRP <5 mg/L and FC <=250 ug/g) at week 112.
Proportion of patients in both treatment arms in endoscopic remission (total SES-CD <5) at week 56 of the study. | Week 56
Proportion of patients in both treatment arms in endoscopic remission (total SES-CD <5) at week 112 of the study | Week 112
Proportion of patients previously enrolled to the ustekinumab 90 mg SC Q8w-arm during REScUE who needed dose optimization to ustekinumab 90 mg SC Q4w at the start or during REScUE-OLE (<=week 100), and that reached endoscopic remission (at week 112. | Week 112
  Proportion of patients previously enrolled to the ustekinumab 90 mg SC Q8w-arm during REScUE who needed dose optimization to ustekinumab 90 mg SC Q4w at the start or during REScUE-OLE (<=week 100), and that reached endoscopic remission (total SES-CD <5) at week 112.
Proportion of patients in both treatment arms in complete endoscopic remission (total SES-CD <3) at week 56 of the study. | Week 56
Proportion of patients in both treatment arms in complete endoscopic remission (total SES-CD <3) at week 112 of the study. | Week 112
Proportion of patients previously enrolled to UST 90 mg SC Q8w-arm during REScUE who needed dose optimization to ustekinumab 90 mg SC Q4w at the start or during REScUE-OLE (<=week 100), and that reached complete endoscopic remission at week 112. | Week 112
  Proportion of patients previously enrolled to the ustekinumab (UST) 90 mg SC Q8w-arm during REScUE who needed dose optimization to ustekinumab 90 mg SC Q4w at the start or during REScUE-OLE (<=week 100), and that reached complete endoscopic remission (total SES-CD <3) at week 112.

OTHER OUTCOMES:
Pharmacokinetic evaluation | between baseline and week 112
  Drug levels in serum
Time until ustekinumab discontinuation (treatment persistence). | between baseline and week 112
Improvements in quality-of-life based on 36-Item Short Form Survey Instrument (SF-36) | between baseline and week 112
  Improvements in quality-of-life based on 36-Item Short Form Survey Instrument (SF-36)
Fatigue as evaluated by the FACIT fatigue scale (functional assessment of chronic illness therapy-fatigue) | between baseline and week 112
  Fatigue as evaluated by the FACIT fatigue scale (functional assessment of chronic illness therapy-fatigue): a 4 point scale, with 0 = not fatigue and 4= very much fatigue
Work productivity as evaluated by the WPAI (work productivity and activity impairment index). | between baseline and week 112
  Work productivity as evaluated by the WPAI (work productivity and activity impairment index).
Pharmaco-economic evaluation | between baseline and week 112
  Pharmaco-economic evaluation of drug cost, hospitalization, work absenteeism, surgery collected and documented during the study

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Pouillon, MD, Principal Investigator — BIRD VZW
Locations (1):
- Ingrid Arijs, Zaventem, Belgium

IPD SHARING:
Plan to Share IPD: No